CLINICAL TRIAL: NCT01631188
Title: Use of Transvenous Pacing Wire During Minimally Invasive Port Access Aortic Valve Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lost nurse researcher support
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Enrique Pantin, Professor, Department of Anesthesiology, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0220110241
Record Dates: First submitted 2012-03-12; First posted 2012-06-29 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Aortic Valve Disease
Keywords: Minimally Invasive Surgery; Port Access Surgery; Heart; Pacing; Wire; MICS; Cardiac Bypass; Epicardial pacing; pacing catheter; pacing wire; pacing swan; pacing pulmonary catheter; Pulmonary Endovent; Catheter; Aortic Valve Surgery; Edwards Lifesciences
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aortic Valve Replacement (Experimental): During surgery your doctor will utilize a new technique using surgical equipment that have already been FDA Approved for other indication. The combination of the equipment and technique will be experimental and will be closely evaluated during and after each case.
  Interventions: Procedure: Minimally Invasive Aortic Valve; Procedure: Minimally Invasive Aortic Valve Surgery; Device: Manipulation in OR surgical technique

INTERVENTIONS:
Procedure: Minimally Invasive Aortic Valve — Patients having minimally invasive aortic valve surgery will have a pacing wire placed through the endovent catheter. The anesthesiologist will attempt to pace the ventricle with this wire if needed to wean from bypass.
Procedure: Minimally Invasive Aortic Valve Surgery — The Anesthesiologist will advance a pacing wire through the Endovent Catheter under TEE in order to pace the heart when the subject is coming off the Cardiopulmonary bypass machine
  Other Names: AVR, Mini AVR, Minimally invasive Port Access Surgery
Device: Manipulation in OR surgical technique — Endovent and pacing wire when coming off cardiopulmonary bypass
  Other Names: AVR, mini avr,

SUMMARY:
The study is being done to determine if the Endovent pulmonary catheter kit, used for port access surgery, can be used as a passageway for a pacing wire. The study hypothesis is that the Endovent kit can be used effectively as a passageway for a pacing wire system.

DETAILED DESCRIPTION:
Many times cardiac surgery requires the use of epicardial pacing in order to wean the patient from bypass. During minimally invasive port access valve surgery, it may not be possible to place the leads on the surface of the heart because of the limited surgical exposure. In this case, transvenous pacing is used. Minimally invasive port access surgery uses specially designed, FDA approved catheters for the procedure. We wish to review the effectiveness of being able to place the wires through the catheters and pace the patient.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age patients having aortic valve port access surgery

Scheduled for Minimally Invasive Port Access Aortic Valve Study

Patient must agree to study participation; understand and sign the written informed consent

Exclusion Criteria:

* < 18 years of age Patients are excluded if they are not having minimaly invasive aortic valve surgery not having aortic valve port access surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique L Pantin, MD, Principal Investigator — Rutgers, The State University of New Jersey; Jonathan Kraidin, MD, Study Director — Rutgers, The State University of New Jersey

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aortic Valve Replacement
Started | 100
Completed | 25
Not Completed | 75
Not completed — Physician Decision | 75

BASELINE CHARACTERISTICS:
Arm/Group | Aortic Valve Replacement
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 74.92 [52 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Were the Endovent Pacing Wire Were Able to Obtain a Ventricular Sensing Signal
Description: Heart to begin pacing upon passing the wire through the catheter to the heart. The catheter would be to be able to pace the heart, with 5 or less milliamps, post heart surgery
Time Frame: Preparing to wean from the cardiopulmonary bypass machine (heart lung machine) until 40 hours post wean.
Population: 23 patients were analyzed. Patient # 12 (male, 75 year) and # 19 (male, 61 year) were eliminated from the study after an intraoperative TEE showed additional pathology that changed the operation needed, and thus the operation from a "mini AVR" to a full sternotomy eliminating the need for the study Endovent pacing lead.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacement
Number analyzed (Participants) | 23
Participants | 23

2. Primary Outcome: Number of Participants That Required Pacing Who Were Able to be Paced
Description: To be able to pace the heart post aortic valve replacement surgery
Time Frame: Preparing to wean from the cardiopulmonary bypass machine (heart lung machine) until 40 hours post wean.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacement
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Number of Participants Who Developed Abnormal Blood Pressure or Heart, and/or Arrhythmias Potentially Related to the Pacing Endovent
Description: Subjects hemodynamic status will be measured and assessed throughout the study including all vital signs
Time Frame: Preparing to wean from the cardiopulmonary bypass machine (heart lung machine) until 40 hours post wean.
Population: 1 of 6 had hemodynamic disturbances significant enough to act immediately. Subject had PVC's, run of wide complex QRS with concurrent drop of systolic blood pressure to 60's, the pacing wire was pulled out of the ventricle, and blood pressure was restored and arrhythmia disappeared.
Measure: Count of Participants; unit: Participants
Arm/Group | Aortic Valve Replacement
Number analyzed (Participants) | 23
Participants
  Participant with arrhythmia not requiring intervention | 5
  Participant with arrhythmia requiring intervention | 1

ADVERSE EVENTS:
Arm/Group | Aortic Valve Replacement
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aortic Valve Replacement (N=23)
hypotension (Cardiac disorders) | 1 — 1 patient of 23 had an episode wide complex QRS vs slow ventricular tachycardia with concurrent drop of systolic blood pressure to 60's that was terminated (arrhythmia and hypotension) by withdrawing the pacing wire back into the Endovent catheter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes